CLINICAL TRIAL: NCT01399294
Title: Traditional Chinese Medicine Syndrome Distribution of Advanced Cancer Patients With Constipation
Brief Title: Cross Sectional Study of Constipation in Advanced Cancer Patients
Status: Completed | Type: Observational
Sponsor: Yan Chai Hospital (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government); Hong Kong Baptist University (Other)
Responsible Party: Dr. Tse Man Wah, Doris / Chief of Service, Department of Medicine & Geriatrics / ICU, Caritas Medical Centre
Other Study IDs: Constipation/TCM2010
Record Dates: First submitted 2011-07-18; First posted 2011-07-21 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Palliative Care; Constipation; Traditional Chinese Medicine
Keywords: Palliative Care; Advanced Cancer; Constipation; Traditional Chinese Medicine; Syndrome Distribution
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Constipation is a common problem in palliative cancer patients. However, there were insufficient randomized controlled trial (RCT) data to identify the "best" laxative or combination of laxatives in these patients.

Traditional Chinese medicine (TCM) in holistic approach is popular among cancer patients. More than half had received at least one form of TCM therapy according to the survey carried in 2008. Chinese herbal medicine (CHM) in compound formulation with nourishing and purging effects simultaneously may be more preferred to relieve constipation by local palliative cancer patients.

TCM syndrome differentiated by collecting all symptoms and signs through the classic four diagnostic methods is the foundation for making diagnosis and prescription in TCM practice.

The present study is the first local study to evaluate the bowel habits and TCM syndrome of advanced cancer patients with constipation. We hope that the results not only can shed light on patient's own reporting or experience of constipation and the effectiveness of current practice, but also can draw up a CHM formulation for advanced cancer patients with constipation.

ELIGIBILITY:
Inclusion Criteria:

* advanced cancer patients
* on medication for facilitating bowel movement and/or constipation visual analogue scale >=2

Exclusion Criteria:

* unable to communicate
* cognitive impaired
* put on colostomy bag
* clinically diagnosed gastrointestinal obstruction
* at end-of-life

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced cancer patients (aged 18 or above) under the care of palliative care units who are on laxatives and who have constipation during recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
TCM syndrome distribution | End of recruitment (estimated timeframe: 3 months)
  Five TCM syndromes, i.e. Excess Heat, Qi Stagnation, Qi Deficiency, Yang Deficiency and Yin Deficiency, are differentiated by TCM practitioner.

SECONDARY OUTCOMES:
bowel habit | End of recruitment (estimated timeframe: 3 months)
  1. Patient's own reporting or experience of constipation
  2. Effectiveness of current practice in relief of constipation

CONTACTS AND LOCATIONS:
Overall Officials: Doris MW Tse, MD, Principal Investigator — Department of Medicine & Geriatrics / ICU, Caritas Medical Centre
Locations (2):
- China (2):
  - Caritas Medical Centre, Hong Kong, Hong Kong
  - Our Lady of Maryknoll Hospital, Hong Kong, Hong Kong